CLINICAL TRIAL: NCT06682338
Title: Psychological Impact of Armed Conflict on Sudanese Diabetic Patients 2024
Status: Completed | Type: Observational
Sponsor: Rayan Jamal Yousif Khidir (Other)
Responsible Party: Sponsor-Investigator, Rayan Jamal Yousif Khidir, Leader of Public Health Group, Research and Publication office
Organization: Research and Publication office (Other)
Other Study IDs: 24004
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Psychological Impact of Armed Conflict; Diabetes Complications
Keywords: DASS-21; Sudan; Psychological; Armed conflict; Diabetics
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study focused on Sudanese people with diabetes who experienced the ongoing war in Sudan. Some people were displaced and others were not. This would had an impact on their mental health. We have investigated this impact and any complications happened to them through Self-Administered questionnaire.

ELIGIBILITY:
Inclusion Criteria: Sudanese Diabetic Patients, both genders, above 18 years

-

Exclusion Criteria:

* Non Diabetic, pre-existing psychological disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sudanese Diabetic Patients above 18 years old, of both genders, from Khartoum and Gezira states.
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2024-04-21 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Psychological Impact | April 2024 - July 2024
  Measured by Depression Anxiety Stress Scale-21 questionnaire.

SECONDARY OUTCOMES:
Diabetes complications | April 2024 - July 2024
  Measured by Self-Administered questionnaire containing questions about demographic data, patient's diabetes history and experienced complications

CONTACTS AND LOCATIONS:
Overall Officials: Alaa MAK Alshykh, BDS, Study Chair — Research and Publication Office, Dental Alumni and Students Affairs, Karary University; Mai AA Balal, BDS, Study Chair — Research and Publication Office, Dental Alumni and Students Affairs, Karary University; Mohamed HA Nasr, PhD, Study Director — International University of Africa / Omdurman Ahlia University; Afaf MH Jabir, BDS, Study Chair — Federal Ministry of Health, Sudan
Locations (1):
- Research and Publication Office, Dental Alumni and Students Affairs, Karary University, Omdurman, Khartoum State, Sudan

IPD SHARING:
Plan to Share IPD: No